CLINICAL TRIAL: NCT03027505
Title: Effectiveness of an Integrated Treatment Protocol for Acute Malnutrition: A Non Inferiority Trial in Passore Province (Northern Region), Burkina Faso
Brief Title: Integrated Treatment Protocol for Acute Malnutrition: A Non Inferiority Trial in Burkina Faso
Acronym: MUAC-Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Association Keoogo (Unknown); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); SOS médecins Burkina Faso (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUAC Only Burkina Faso
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Global Acute Malnutrition (GAM)
Keywords: MUAC; Acute malnutrition; RUTF; Children; Burkina Faso

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MUAC<125mm (Experimental): no medical complication
  Interventions: Drug: Ready to Use Therapeutic Food (RUTF)

INTERVENTIONS:
Drug: Ready to Use Therapeutic Food (RUTF) — MUAC used as the primary admission and exit criteria for children with MUAC <125mm and no medical complication.
  Single treatment of RUTF for severe and moderate malnourished children and gradual reduction of doses according to the MUAC and the weight of the child during treatment. MUAC split into 3 categories:
  * MUAC <115 mm: 175 kcal /kg/day
  * 115 <MUAC <120mm: 125kcal/kg/day
  * 120 <MUAC <125mm: 75kcal/kg/day
  Other Names: MUAC<125mm

SUMMARY:
MUAC only is a pilot trial external control carried out between January 2017 and December 2017 in the Yako district (northern region), Burkina Faso.

The objective of this study is to evaluate an integrated protocol for acute malnourished children without medical complication. The hypotheses of the integrated protocol include :

1. A global treatment of acute malnutrition (moderate and severe) with a single treatment (RUTF) would improve the functioning of the program through early identification of acutely malnourished children, while achieving a better coverage and using a single supply chain.
2. A gradual reduction of RUTF dosage according to a child's MUAC status could significantly increase the number of children on treatment without increasing overall RUTF quantity while maintaining similar recovery rates.

DETAILED DESCRIPTION:
Objectives :

Main objective :

To ensure the recovery rate of the integrated protocol for treatment of acute malnutrition is significantly greater than 75% (reference value of the national program in BF).

Secondary objectives :

* To ensure the mortality rate of the integrated protocol for treatment of acute malnutrition is significantly lower than 3% (reference value of the national BF program).
* To ensure the default rate of the integrated protocol for treatment of acute malnutrition is significantly lower than 15% (reference value of the national BF program).
* To ensure the non-response rate of the integrated protocol for treatment of acute malnutrition is significantly lower than 8%.
* To ensure the hospitalization rate of the integrated protocol for treatment of acute malnutrition is significantly lower than 15%.
* To ensure the coverage rate of the program increases by 30% after the year the integrated protocol was introduced (specific protocol annexed).
* To estimate the relapse rate of the integrated protocol for treatment of acute malnutrition.
* To compare RUTF rations per child of the integrated protocol compared to the national protocol

Methods :

The study population will include all acutely malnourished children aged between 6 and 59 months seeking consultations at all of the health centers in Yako District between January 2017 and December 2017.

The study will be implemented in Burkina Faso's Yako District, which includes 54 health centers.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6 and 59 months old
* New admission
* Acute malnutrition defined as follows:

  * MUAC<125mm
  * MUAC> 125mm AND WHZ (Z-score) <-3 (WHO standard)
  * Edema
* Resident in the study area (Yako district)
* Signed informed consent of the mother or the child's guardian

Exclusion Criteria:

* Children allergic to milk, peanuts and / or RUTF

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4958 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Recovery rate | Between 4 and 12 weeks
  The recovery is defined as below :
  * Minimum of 4 weeks of participation in the program
  * MUAC> = 125 mm on 2 consecutive visits
  * No edema for minimum 2 weeks
  * Good Clinical Health

SECONDARY OUTCOMES:
Mortality rate | Between inclusion and week 12
Default rate | Between 3 and 12 weeks
  Patient absent for 3 consecutive visits
Non-respondent rate | 12 weeks after inclusion
  Patient who not reach the recovery criteria after twelve weeks in the program
Hospitalization rate | Between inclusion and week 12
Relapse rate | up to 3 months
  Patient having reached the recovery criteria and returning for a new episode of malnutrition (MUAC<125mm).
  The children's MUAC will be measured at home 3 months after program exit. For organizational and financial reasons, this data will not be collected for all children. A specific protocol explaining the sampling and organization of data collection will be annexed to the protocol.
RUTF rations | Between inclusion and week 12
  Total number of RUTF bags received per child during participation in the program.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shepherd, MD, Principal Investigator — Directrice de recherches Opérationnelles et Médicales, ALIMA, USA; Renaud Becquet, MPH,PhD,HDR, Principal Investigator — Chercheur Inserm, Inserm U1219 Bordeaux Population Health Center-Université de Bordeaux
Locations (1):
- ALIMA, Yako, Nord Region, Burkina Faso

IPD SHARING:
Plan to Share IPD: No